CLINICAL TRIAL: NCT04567563
Title: The Physiological Effects of Remote Ischemic Conditioning on the Healing of Diabetic Foot Ulcers
Brief Title: Remote Ischemic Conditioning and Diabetic Foot Ulcers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Des Moines University (Other)
Collaborators: Iowa State University (Other)
Responsible Party: Principal Investigator, Katherine Frush, Associate Professor, Des Moines University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-2020-3
Record Dates: First submitted 2020-09-17; First posted 2020-09-28 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Diabetic Foot Ulcer; Diabetic Angiopathies
Keywords: remote ischemic conditioning; diabetic foot ulcer; diabetic angiopathy
MeSH Terms: conditions — Diabetic Foot; Diabetic Angiopathies

STUDY DESIGN:
Intervention Model Description: Will have intervention group and standard of care group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote Ischemic Condition (Active Comparator)
  Interventions: Device: Remote Ischemic conditioning (RIC)
- Standard of Care (No Intervention)

INTERVENTIONS:
Device: Remote Ischemic conditioning (RIC) — Intervention Group: Patients will self-administer RIC treatment with the LifeCuff device 3 times a week. Treatment will be delivered at the patient's home and compliance will be monitored by the LifeCuff device. Control Group: Patients undergo typical standard of care treatment. Assessment of Ulcer Closure: Ulcers will be assessed as completely closed by the Principal Investigator through clinical judgement and photographic support. Patients that completely heal their ulcer during the healing period will complete the study and no further blood or tissue measurements will be taken
  Arms: Remote Ischemic Condition

SUMMARY:
Study type: Randomized, double blinded, interventional, single-site study. Two groups: Active receiving RIC therapy from the LifeCuff device and standard of care treatment without RIC.

Study population: Adults (18 to 90) with diabetes myelitis presenting with diabetic foot ulcers.

Randomization and sample size: Subjects will be allocated on a 1:1 ratio, yielding a minimum per protocol population (PP Population) of 15 patients in the Active group and 15 in the control group.

Study timeline: Total amount of time from the Screening Visit to the Final Visit is approximately 16 weeks. For patients who meet inclusion criteria, they are randomized into Active or Control treatment groups. In addition they are stratified into groups based on wound etiology: neuropathic (defined as insensate at 2 or more of 5 sites verified by insensitivity to the 5.07 Semmes-Weinstein 10 g monofilament), ischemic (defined as ABI of 0.7 neuro-ischemic (meeting both of above criteria) Subjects will present at DMU Foot and Ankle Clinic on weeks 0, 3, 6, 9, and 12 for the following measurements: 40mL venous blood draw (VEGF, SDF1a) 2mm punch biopsy (CD34+) Local wound perfusion (Laser Speckle[FK2] ) Ulcer size measured by digital planimetry (TissueAnalytics)

ELIGIBILITY:
Inclusion Criteria:

* Patient any gender between the ages of 18 and under 90 at the time of consent.
* Target ulcer has a minimum area of 1.0 cm2 and a maximum area of 20.0 cm2, measured at screening after sharp debridement, as assessed by computerized planimetry.
* Target ulcer open for a minimum of 4 weeks and a maximum of 52 weeks duration prior to the screening visit.
* Target ulcer is located on the toe or lateral dorsal, or plantar aspect of the foot with no portion on the ankle.
* Target ulcer is Grade IC (ischemic, non-infected superficial wound) or IIC (ischemic non-infected wound penetrating to tendon or capsule), according to the University of Texas Diabetic Wound Classification system.
* Adequate perfusion without critical limb ischemia, confirmed by vascular assessment of the affected foot through any of the following methods: ABI >0.7
* Confirmed diagnosis of type 1 or 2 diabetes mellitus
* Patient has a glycated hemoglobin A1c (HbA1c) level of less than 12%
* If patient has two or more ulcers, they must be separated by at least 2 cm and the largest one will be included as the study DFU though all will be similarly treated
* Patient is willing to use prescribed off-loading method during the whole duration of the study
* Patient available for the entire study period all follow up visit requirements, and able and willing to adhere to protocol requirements
* Patient able and willing to give written informed consent

Exclusion Criteria:

* Target ulcer is less than 1.0 cm2 measured at consent after sharp debridement
* Target ulcer is due to a non-diabetic etiology
* Presence in target ulcer of cellulitis, osteomyelitis or other clinical evidence of infection at time of enrollment.
* Presence of any foot ulcer (whether or not on the target foot) for which systemic antibiotic treatment is required.
* A history of more than 8 weeks' treatment with immunosuppressants (including systemic corticosteroids), cytotoxic chemotherapy, or application of topical steroids to the ulcer surface within one month prior to initial screening, or treatments with such medications during the screening period.
* Patients with an amputation on the affected foot, if it impedes proper offloading of the target DFU.
* Patients with active Charcot foot, or inactive Charcot foot, if it impedes proper offloading of the target DFU.
* Women who are pregnant or considering becoming pregnant within the next 6 months.
* Patients with concurrent severe psychiatric disease that in the opinion of the investigator would impede participation in the trial.
* Presence of subject having recent or current alcohol or drug abuse.
* Patients with severe kidney disease who are currently untreated or awaiting dialysis treatment
* Participation in another study involving treatment with an investigational product within the previous 30 days.
* Any other medical or psychological conditions that, in the opinion of the Investigator may make patient's participation unreliable or may interfere with study assessments.
* Patients with history of radiation to the ulcer

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-11 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Change in ulcer area and overall healing rate | will be evaluated at 0, 3, 6, 9 and 12 weeks
  Will evaluate healing rates and times for both treatment group and standard of care group using app that can take picture and measure area

SECONDARY OUTCOMES:
VEGF | will be evaluated at 0, 3, 6, 9 and 12 weeks
  Will evaluate blood levels of VEGF in treatment group and standard of care group
SDF1a | will be evaluated at 0, 3, 6, 9 and 12 weeks
  Will evaluate blood levels of SDF1a in treatment group and standard of care group
CD34+ | will be evaluated at 0, 3, 6, 9 and 12 weeks
  Will evaluate soft tissue biopsy for presence or absence of CD34+ in treatment group and standard of care group
tissue perfusion | will be evaluated at 0, 3, 6, 9 and 12 weeks
  Will evaluate overall tissue perfusion using Laser Speckle imaging for both treatment group and standard of care group

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Frush, DPM, Principal Investigator — Des Moines University

IPD SHARING:
Plan to Share IPD: No